CLINICAL TRIAL: NCT02185924
Title: COMBINATION OF CONTINUOUS FEMORAL BLOCK AND INTRAVENOUS PARECOXIB FOR POSTOPERATIVE ANALGESIA AFTER TOTAL KNEE ARTHROPLASTY. A DOUBLE BLIND PROSPECTIVE STUDY.
Brief Title: Combination of Continuous Femoral Block and Intravenous Parecoxib For Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Despoina Sarridou, ANAESTHESIOLOGIST, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: S-138/15-06-10
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: POSTOPERATIVE ANALGESIA FOR TKA PARECOXIB/CFB
Keywords: PARECOXIB; CONTINUOUS FEMORAL BLOCK
MeSH Terms: interventions — parecoxib; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTINUOUS FEMORAL BLOCK AND PARECOXIB (Experimental): Continuous infusion of0,2% of ropivacaine at 10 ml/h and 2 mls (40 mg) of iv parecoxib
  Interventions: Drug: Parecoxib; Drug: CONTINUOUS FEMORAL BLOCK WITH ROPIVACAINE 0,2%
- CONTINUOUS FEMORAL BLOCK AND PLACEBO (Placebo Comparator): Continuous infusion of 0.2% ropivacaine at 10 ml/h and 2 mls of iv N/S0.9%
  Interventions: Drug: CONTINUOUS FEMORAL BLOCK WITH ROPIVACAINE 0,2%; Drug: N/S 0.9%

INTERVENTIONS:
Drug: Parecoxib
  Other Names: DYNASTAT
  Arms: CONTINUOUS FEMORAL BLOCK AND PARECOXIB
Drug: CONTINUOUS FEMORAL BLOCK WITH ROPIVACAINE 0,2%
  Other Names: NAROPEINE
Drug: N/S 0.9%
  Other Names: PLACEBO
  Arms: CONTINUOUS FEMORAL BLOCK AND PLACEBO

SUMMARY:
Combination of continuous femoral block with parEcoxib vs placebo. Investigation of morphine consumption, opioid sparing effects, VAS pain scores, haemodynamics, Anxierty scores, transfusion requirements , Range of motion and rehabilitation parameters between two groups

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS ASA I-II UNDERGOING TOTAL KNEE ATRTHROPLASTY

Exclusion Criteria:

Exclusion criteria for both groups included:

* Age younger than 40 years old or older than 80 years old
* ASA > III
* Obesity (>140 kg body weight)
* Allergy to local anesthetics
* History dependence on opioids
* Contraindications for subarachnoid anesthesia or femoral block (coagulopathy, local infection, pre-existing neurological problems, patient refusal)
* Contraindications to the administration of parecoxib
* Severe hepatic or renal disease (serum creatinine ≥ 1.7 mg/dl)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
MORPHINE CONSUMPTION WITH PCA BETWEEN TWO GROUPS | 36/h POSTOPERATIVELY
VAS PAIN SCORES BETWEEN TWO GROUPS | 36/h POSTOPERATIVELY
HAEMODYNAMIC PARAMETERS BETWEEN TWO GROUPS | During perioperative period

SECONDARY OUTCOMES:
ANXIETY LEVELS | 36 HOURS POSTOPERATIVELY
  ANXIETY SCORES WERE QUANTIFIED USING THE SPIELBERG INVENTORY

OTHER OUTCOMES:
RANGE OF MOTION, TRANSFUSION REQUIREMENTS, VAS SCORES POSTOPERATIVELY | AFTER 36 HOURS POSTOPERATIVELY
MODIFIED BROMAGE SCALE | 36/h POSTOPEPATIVELY

CONTACTS AND LOCATIONS:
Overall Officials: DESPOINA SARRIDOU, SENIOR REGISTRAR, Principal Investigator — SENIOR CLINICAL FELLOW THE ROYAL BROMPTON AND HAREFIELD TRUST, SENIOR REGISTRAR IN ANAESTHESIA ASKLEPEION VOULAS
Locations (1):
- Department of Anaesthesia Asklepeion Voulas General Hospital, Voula Athens, Greece

REFERENCES:
- [Derived] Sarridou DG, Chalmouki G, Braoudaki M, Siafaka I, Asmatzi C, Vadalouka A. Parecoxib Possesses Anxiolytic Properties in Patients Undergoing Total Knee Arthroplasty: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Clinical Study. Pain Ther. 2016 Jun;5(1):55-62. doi: 10.1007/s40122-016-0046-1. Epub 2016 Feb 9. PMID 26861666